CLINICAL TRIAL: NCT06279650
Title: Self-hypnosis Training in Chronic Pain Management: A Qualitative Exploratory Study of Patients Practicing Self-hypnosis
Brief Title: Self-hypnosis Training for Chronic Pain Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, David Ogez, Clinical Assistant Professor, Department of Anesthesiology and Pain Medicine, Université de Montréal, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-2741
Record Dates: First submitted 2024-02-01; First posted 2024-02-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypnosis, Chronic Pain Management
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-hypnosis (Experimental)
  Interventions: Other: Self-hypnosis
- Psyco-education and cognitive behavioral therapy (Active Comparator)
  Interventions: Other: Psycho-education and cognitive Bahavioral therapy (CBT)

INTERVENTIONS:
Other: Self-hypnosis — The HYlaDo intervention comprises 8 90-minute sessions. Session 1 offers psycho-education on pain and medical hypnosis. Sessions 2 to 7 offer brief introductions followed by hypnosis induction, during which the CBT elements (exposure and cognitive restructuring) to be worked on during the session are introduced. The sessions are aimed at managing: 2- anxiety and mood; 3- pain dramatization; 4- and 5- pain perception; 6- kinesiophobia; 7- future projection and resource mobilization. Session 8 provides feedback and recommendations for independent practice. Each hypnosis follows the same pattern: induction, deepening, CBT-based hypnotic work, post-hypnotic suggestions and return to wakefulness, explanations of the exercise and recommendations for independent practice.
  Arms: Self-hypnosis
Other: Psycho-education and cognitive Bahavioral therapy (CBT) — The psychoeducation-CBT intervention for pain and anxiety/depression consists of 8 90-minute sessions. It has already been implemented in HMR's pain clinic, and controls both the effects of time and repetition of measures, as well as non-specific factors including expectations associated with receiving active treatment, therapeutic relationship, frequency of encounters, and participation in a manualized intervention. It is designed to inform participants about pain, its costs, neurophysiology, nature and impact. It includes general information on pain, as well as information tailored to the participants' particular type of pain. The sessions are interactive, with the therapist stimulating discussion of the educational content and its relevance to the participants' lives.
  Arms: Psyco-education and cognitive behavioral therapy

SUMMARY:
Title: Self-hypnosis training in chronic pain management: A pilot study Our primary objective concerns the effect of hypnosis intervention on change in 24h pain between T0 (pre-intervention) and T4 (3-month follow-up). The secondary objectives concern the effects of the intervention on (i) change in 24h pain between T0 and T5 (6-month follow-up), (ii) changes from T0 in measures of the functional impact of pain, (iii) changes from T0 in anxiety-depression scores and (iv) changes from T0 in quality of life.

The study design is a Randomized efficacy pilot study. The study focuses on patients practicing self-hypnosis within HMR groups. The study population is pain clinic patients. The sample size is 60 pain clinic patients. Study duration: February 2024 - December 2024. Center responsible for the study: Centre de Recherche de l'Hôpital Maisonneuve-Rosemont (CR-HMR) - CEMTL, Montreal, Quebec, Canada.

Adverse events: none expected.

DETAILED DESCRIPTION:
A self-hypnosis training program has been developed based on the experience of the program developed in medical oncology (phase I). The aim of this project is to analyze the self-hypnosis practice of chronic pain patients, and to evaluate the training program provided in pain management clinics, by means of qualitative research interviews. It is therefore situated at level Ib of the ORBIT model: Program refinement. Through this study, the investigators also wish to evaluate the effects of the intervention on users. In this context, the investigators hypothesize that patients who practice self-hypnosis show an improvement in their quality of life and a reduction in anxiety and pain levels. At this level, there are two objectives :

1. To assess the effect of hypnosis intervention on change in 24h pain between T0 (pre-intervention) and T3 (3-month follow-up).
2. To assess the effects of hypnosis intervention on (i) change in 24h pain between T0 and T4 (6-month follow-up), (ii) changes from T0 in measures of the functional impact of pain, (iii) changes from T0 in anxiety-depression scores and (iv) changes from T0 in quality of life.

Methods

Intervention : Self-hypnosis training Based on the exercises from the oncology pilot project, the investigators redefined a program applicable to the pain clinic (phase I ORBIT). To do so, the investigators maintained the stress and pain management exercises and removed the exercises relating to the management of secondary symptoms of cancer treatment. This new self-hypnosis training program is based on four complementary exercises: two on stress management and two on pain perception. Each exercise is organized according to the same hypnotic framework: induction, deepening, hypnotic work, post-hypnotic suggestions and return to the waking state. Each exercise is derived from the oncology study and has been enhanced by protocols drawn from the experience of other hypnotherapists.

The first exercise involves letting go of the emotions and stress associated with the painful condition, using the rucksack technique: a metaphor enabling the patient to empty an imaginary bag that is heavy and preventing him or her from moving forward. The weight of the bag represents the negative emotions, losses and pain that weigh down the patient's daily life. The second exercise focuses on the notion of acceptance, in the same way as cognitive-behavioral acceptance therapies. Suggestions and metaphors used in the work include the ideas of doing nothing, letting oneself be carried away and meditating in a pleasant place. The third exercise uses visualization techniques to modify pain. The modification concerns the form and intensity of the pain. Finally, the fourth exercise is derived from Rossi's protocol, which proposes mobilizing the patient's resources through levitation and catalepsy techniques. This technique focuses on the body and aims to restore confidence in the body in people with pain.

Participants: Sixty participants from pain clinic of our institution will be included in these research. They will be randomized in the two group of our study : hypnosis Vs Psychoeducation/CBT.

Procedures: Five measurement times will be used: T1-Start of research project; T2 - Mi-intervention, T3 - End of intervention, T4 - 3 months follow up, T5 - 6 months follow up. At each of these times, participants will complete self-administered questionnaires (pain, anxiety-depression and quality of life). The investigators will also collect a self-hypnosis practice diary, which the patient will complete during the course of the study: each week, the patient will note each practice in his or her diary, indicating the time and duration of the practice.

Measures: 24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine). The functional impact of pain will be measured using the Brief Pain Inventory (BPI). This 9-item scale assesses (1) the presence of pain, (2) the location of the pain, (3) the most intense pain, (4) the least intense pain, (5) the pain felt in general, (6) the pain felt at the moment on a NRS of 0 to 10. It also documents (7) the treatments used and (8) the relief provided over the last 24 hours. Item (9) concerns a subscale that documents the extent to which pain has interfered with 7 different activity and response domains (e.g., general activity, mood, relationships with others) over the last 24 hours, using an NRS from 0 to 10 (0 = pain does not interfere with this activity, 10 = pain interferes completely).

Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS). This scale was developed for general practice patients and comprises 2 subscales of 7 items each, measuring anxiety and depression respectively. Each item is scored between 0 and 3. The score of each subscale is obtained by summing the scores of the 7 items, with a total score thus ranging from 0 to 21. The scale has been translated and validated in French.

Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains: (1) Limitations in physical activities due to health problems; (2) Limitations in social activities due to physical or emotional problems; (3) Limitations in usual activities due to physical health problems; (4) Body pain; (5) General mental health (psychological distress and well-being); (6) Limitations in usual activities due to emotional problems; (7) Vitality (energy and fatigue); (8) General perception of health. The scores for the various domains are converted and pooled using a scoring key, to obtain a total score indicating a range of quality of life from low to high. Two component scores can also be tallied: a summary of the physical component and a summary of the mental component. Secondary measures concern hypnosis practice. The level of practice will be collected from the logbook. Participants will also be asked to self-assess their perceived levels of relaxation using a VAS-10 scale (0 = "not at all relaxed"; 10 = "very relaxed") before and after practice.

Analyses: Primary and secondary outcome measures will be compared across the three time points using repeated measures ANOVAs, and effect sizes will be calculated to document changes associated with the intervention. The investigators will also conduct correlations between self-hypnosis practice and scores on the measures taken. The investigators expect to see relationships between significant levels of practice and improvements in quality of life, and reductions in anxiety and pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were to have participated in the past year in the self-hypnosis training program and to agree to take part in these research interviews.
* be 18 years of age or older;
* have received one of the above diagnoses, confirmed by medical record review or physician confirmation;
* report pain that has been present for at least 3 months;
* have a pain intensity over the last 24 hours (24h pain) of at least 4 on a Numerical Rating Scale (NRS) from 0 to 10 at baseline;
* be able to read, speak and understand French;
* have Internet access and be able to participate in a telepractice intervention group and complete online questionnaires.

Exclusion Criteria:

* have deafness and/or severe cognitive impairment that may impair communication;
* have current or recent psychiatric instability (e.g., active suicidal ideation, active delusional or psychotic thoughts) that could interfere with participation, as assessed by a clinical psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time 1 : Numerical Rating Scale (NRS) from 0 to 10 | First day
  24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine)
Time 1 : Questionnaire Brief Pain Inventory (BPI) | First day
  The functional impact of pain will be measured using the Brief Pain Inventory (BPI) with 9-item scale assesses.
Time 1 : Hospital anxiety and depression scale (HADS) | First day
  Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS).
Time 1 : SF-36 (36-Item Short Form Survey) | First day
  Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.
Time 1 : Questionnaire socio-demographic and clinical | First day
  A socio-demographic and clinical questionnaire will also be requested.

SECONDARY OUTCOMES:
Time 2 : Numerical Rating Scale (NRS) from 0 to 10 | 1 month
  24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine).
Time 2 : Questionnaire Brief Pain Inventory (BPI) | 1 month
  The functional impact of pain will be measured using the Brief Pain Inventory (BPI) with 9-item scale assesses.
Time 2 : Hospital anxiety and depression scale (HADS) | 1 month
  Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS).
Time 2 : SF-36 (36-Item Short Form Survey) | 1 month
  Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.

OTHER OUTCOMES:
Time 3 : Numerical Rating Scale (NRS) from 0 to 10 | 2 months
  24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine).
Time 3 : Questionnaire Brief Pain Inventory (BPI) | 2 months
  The functional impact of pain will be measured using the Brief Pain Inventory (BPI) with 9-item scale assesses.
Time 3 : Hospital anxiety and depression scale (HADS) | 2 months
  Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS). Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.
Time 3 : SF-36 (36-Item Short Form Survey) | 2 months
  Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.
Time 4 : Numerical Rating Scale (NRS) from 0 to 10 | 3 months
  24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine).
Time 4 : Questionnaire Brief Pain Inventory (BPI) | 3 months
  The functional impact of pain will be measured using the Brief Pain Inventory (BPI) with 9-item scale assesses.
Time 4 : Hospital anxiety and depression scale (HADS) | 3 months
  Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS).
Time 4 : SF-36 (36-Item Short Form Survey) | 3 months
  Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.
Time 5 : Numerical Rating Scale (NRS) from 0 to 10 | 6 months
  24 h pain will be measured using the NRS from 0 to 10 (0 = no pain, 10 = the most horrible pain participants can imagine).
Time 5 : Questionnaire Brief Pain Inventory (BPI) | 6 months
  The functional impact of pain will be measured using the Brief Pain Inventory (BPI) with 9-item scale assesses.
Time 5 : Hospital anxiety and depression scale (HADS) | 6 months
  Anxiety-depression will be assessed using the Hospital anxiety and depression scale (HADS).
Time 5 : SF-36 (36-Item Short Form Survey) | 6 months
  Quality of life will be assessed by the SF-36 (36-Item Short Form Survey), which comprises 36 questions covering eight health domains.

CONTACTS AND LOCATIONS:
Locations (1):
- 5415 Bd de l'Assomption, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided